CLINICAL TRIAL: NCT06241404
Title: Efficacy of Therapeutic Exercise vs. Treatment of Myofascial Trigger Points in Shoulder Tendinopathies: Randomised Clinical Trial
Brief Title: Efficacy of Therapeutic Exercise vs. Treatment of Myofascial Trigger Points.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 250124
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Tendinopathy
Keywords: shoulder tendinopathy; supraspinatus; infraspinatus; physiotherapy techniques; therapeutic exercise; trigger points
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic exercise group (Experimental): patients who have been treated for shoulder tendinopathy by exercise therapy
  Interventions: Procedure: Exercise therapy
- trigger points group (Active Comparator): patients who have been treated for shoulder tendinopathy by trigger point therapy
  Interventions: Procedure: trigger point therapy

INTERVENTIONS:
Procedure: trigger point therapy — patients who have been treated for shoulder tendinopathy by trigger point therapy
  Arms: trigger points group
Procedure: Exercise therapy — patients who have been treated for shoulder tendinopathy by exercise therapy
  Arms: therapeutic exercise group

SUMMARY:
Background: Shoulder pain commonly affects the general population, with rotator cuff tendinopathy being the most common cause.

the most common cause, with rotator cuff tendinopathy diminishing function and quality of life, leading to a major socio-economic impact.

quality of life, leading to a major socio-economic impact. As a result, there are two treatment approaches with potential effectiveness: therapeutic exercise (TE) and myofascial trigger point treatment (TMT).

trigger point treatment (TTP).

Objective: The main objective of this randomised clinical trial is to determine the efficacy of ET versus treatment of MTPs in shoulder tendinopathies.

Methods: For this study, 20 participants were randomly divided into two groups: a ET group, with which a 10-exercise programme was initiated (n = 10), and a PGM group which was given an intervention protocol (n = 10).

intervention protocol (n = 10). Both received a total of 10 sessions. Pain intensity pain intensity, pressure pain threshold (PPT) and range of motion (ROM) were assessed before starting and after 10 sessions.

and after 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Patients diagnosed by an orthopaedic surgeon with shoulder tendinopathy. tendinopathy.
* Symptoms of shoulder pain lasting more than 3 months.
* Pain on Jobe, Patte and infraspinatus assessment manoeuvres (highlighting abduction and abduction and external rotation).

Exclusion Criteria:

* Previous shoulder surgery.
* Radiating (non-referred) pain from cervical radiculopathy.
* Shoulder pain associated with other diagnoses (Examples: retractile capsulitis, subacromial syndrome, tendon rupture, posterosuperior conflict, etc.).

subacromial syndrome, tendon rupture, posterosuperior conflict, etc).

* Patients with multiple pathologies.
* Patients with neurological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Range of motion | At the end of Session 10 (each Session is 7 days)
  measurement of shoulder range of motion
pain intensity | At the end of Session 10 (each Session is 7 days)
  measured on a VAS scale where 0 is the minimum and 10 is the maximum.

SECONDARY OUTCOMES:
pressure pain threshold | At the end of Session 10 (each Session is 7 days)
  measured by algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Velázquez Saornil, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoma M, Herrington L, Mackenzie TA. The Effect of Exercise Therapy Interventions on Shoulder Pain and Musculoskeletal Risk Factors for Shoulder Pain in Competitive Swimmers: A Scoping Review. J Sport Rehabil. 2022 Feb 23;31(5):617-628. doi: 10.1123/jsr.2021-0403. Print 2022 Jul 1. PMID 35196648
- [Background] Jung KM, Choi JD. The Effects of Active Shoulder Exercise with a Sling Suspension System on Shoulder Subluxation, Proprioception, and Upper Extremity Function in Patients with Acute Stroke. Med Sci Monit. 2019 Jun 30;25:4849-4855. doi: 10.12659/MSM.915277. PMID 31256191
- [Background] Spanhove V, De Wandele I, Malfait F, Calders P, Cools A. Home-based exercise therapy for treating shoulder instability in patients with hypermobile Ehlers-Danlos syndrome/hypermobility spectrum disorders. A randomized trial. Disabil Rehabil. 2023 Jun;45(11):1811-1821. doi: 10.1080/09638288.2022.2076932. Epub 2022 May 24. PMID 35609204
- [Background] Richmond H, Lait C, Srikesavan C, Williamson E, Moser J, Newman M, Betteley L, Fordham B, Rees S, Lamb SE, Bruce J; PROSPER Study Group. Development of an exercise intervention for the prevention of musculoskeletal shoulder problems after breast cancer treatment: the prevention of shoulder problems trial (UK PROSPER). BMC Health Serv Res. 2018 Jun 18;18(1):463. doi: 10.1186/s12913-018-3280-x. PMID 29914494
- [Background] Lin IH, Chang KH, Liou TH, Tsou CM, Huang YC. Progressive shoulder-neck exercise on cervical muscle functions in middle-aged and senior patients with chronic neck pain. Eur J Phys Rehabil Med. 2018 Feb;54(1):13-21. doi: 10.23736/S1973-9087.17.04658-5. Epub 2017 Jul 17. PMID 28714658
- [Result] Fathollahnejad K, Letafatkar A, Hadadnezhad M. The effect of manual therapy and stabilizing exercises on forward head and rounded shoulder postures: a six-week intervention with a one-month follow-up study. BMC Musculoskelet Disord. 2019 Feb 18;20(1):86. doi: 10.1186/s12891-019-2438-y. PMID 30777064
- [Result] Eshoj H, Rasmussen S, Frich LH, Hvass I, Christensen R, Jensen SL, Sondergaard J, Sogaard K, Juul-Kristensen B. A neuromuscular exercise programme versus standard care for patients with traumatic anterior shoulder instability: study protocol for a randomised controlled trial (the SINEX study). Trials. 2017 Feb 28;18(1):90. doi: 10.1186/s13063-017-1830-x. PMID 28245853
- [Derived] Villa Munoz T, Velazquez Saornil J, Sanchez Mila Z, Romero-Morales C, Almazan Polo J, Baraja Vegas L, Hugo-Villafane J, Abuin-Porras V. Comparative evaluation of the efficacy of therapeutic exercise versus myofascial trigger point therapy in the treatment of shoulder tendinopathies: a randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Oct 16;10(4):e002043. doi: 10.1136/bmjsem-2024-002043. eCollection 2024. PMID 39430399